CLINICAL TRIAL: NCT04045119
Title: Effect of a Facial Cream Containing 0.5% Cannabidiol and 0.1% Hemp Oil on Skin Hydration and Characteristics Associated Acne-prone Skin
Brief Title: Effect of a Facial Cream Containing Cannabidiol and Hemp Oil on Skin Hydration and Acne-prone Skin
Acronym: Dahlia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avicanna Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Av 0002 DaCol
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cosmetic Acne
Keywords: CBD; Cosmetics; Acne-prone skin; Oily Skin

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental (i.e., prospective, non-randomized, non-controlled), open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before-and-after (Experimental): 54 Healthy adults 18 years of age or older at the visit or will receive the first application and will be evaluated according to the objectives defined in the study (short-term data) and to evaluate the longterm effects, two other visits will be made at intervals of 2 weeks to evaluate the impact of topical skin application according to the parameters defined in the study
  Interventions: Other: Topical Moisturizer

INTERVENTIONS:
Other: Topical Moisturizer — The investigational product is a moisturizing facial cream for skin with imperfections that is applied topically and is manufactured by Avicanna Inc. This preparation contains widely used ingredients from mineral and botanical origin aimed at improving skin hydration and characteristics associated acne-prone skin. The moisturizer also contains 0.1% of hemp oil rich in essential fatty acids and antioxidants and 0.5% of cannabidiol with regulatory effect on the skin.

SUMMARY:
This research seeks to evaluate the short (i.e., after single application) and long-term (i.e., after periodic application) hydrating effect of a topical preparation containing CBD and hemp oil on facial skin as well as the effect on erythema, appearance, instrumentally measured sebum production and quality of life.

DETAILED DESCRIPTION:
In this research effort, hypothesis is that application of the topical product improves skin hydration as measured instrumentally by its electric properties as well as other variables associated with skin hydration, sebum production and appearance. Therefore, this research effort seeks to evaluate the short (i.e., after single application) and long-term (i.e., after periodic application) hydrating effect of a topical preparation containing CBD, rosemary extract and hemp oil on facial skin. For this purpose, objective measures aimed at stablishing the change of parameters related to skin water content will be measured. Additionally, other measurements will be obtained to establish the change of different parameters related to the effect on appearance, instrumentally measured sebum production and quality of life. These include: instrumental and subjective measurement of oily skin and standardized photography for assessment of imperfections as well as, a validated assessment of the impact of acne-prone skin on quality of life.

Healthy adults will be invited to participate and the general characteristics of the product will be explained, as well as the amount of time that will be required. The individuals that agree to participate will have to read and sign the informed consent, register contact information, and will be scheduled for visit 0 at the research center within 2 to 7 days. During this period (i.e., washout period), the subject will be told not to use abrasive cleansing products or topical medicines on the facial skin, not to take more than one shower per day, and not to consume caffeine or alcohol 24 hours before attending the research center.

During the washout period the subject will receive a call to confirm compliance with washout requirements as well as visit 0 schedule. If washout conditions are not met, subject will be reminded to comply and visit will be re-scheduled within 2 to 7 days.

In visit 0 at the research center, contact information, demographic variables and standard anthropometric variables will be recorded. Subsequently, the subject will be given detailed information about the research product and protocol, accompanied by an information leaflet with indications regarding the use of the investigational product as well as recommendations on preferred hygiene regimens.

The subject will be able to review the material in a room under controlled ventilation, temperature, humidity and lighting conditions, where he or she will have to stay for a minimum of 30 minutes. After that, in an adjacent room under the same conditions, the basal characteristics of the facial skin will be measured through electrical and photometric variables as well as self-assessment of oily skin, a standardized photograph with visual assessment and self-image questionnaire (i.e., hour 0). The bioengineering measurements will be made on the cheeks (i.e., between the base of the ear lobe and the apex of the chin) and forehead (i.e., exact center of the forehead) and no marking of the measurement area will be performed.

Once this process is done, the subject goes back to the waiting room, where a research assistant explains how to apply the investigational product on the face and evaluate the product characteristics. The subject applies the product and evaluates its characteristics. 10 minutes after application, the subject will complete a perception survey about the product characteristics sensation produced on the skin. Afterwards, the subject may leave the room under controlled conditions; however, he or she must return 30 minutes prior to the next measurements.

One hour after the application of the topical product (including 30 minutes of acclimatization in the room under controlled conditions), a new measurement of the electrical, photometric and colorimetric variables as well as self-assessment of oily skin and a standardized photograph with visual assessment is made. This procedure is repeated after 3 hours (including 30 minutes of acclimatization in the room under controlled conditions). Once the last measurement is made the subject completes the last part of the survey and is given a vessel containing the investigational product and instructions regarding its usage will be reinforced. Additionally, schedule for next visit will be determined at this time.

The subject must apply the product according to the indications and keep a journal of the applications. Additionally, the subject must refrain from using other topical products on the volar forearm or systemic products that may alter the skin conditions. Furthermore, there will be a follow-up call to remind the participant to comply with the requirements and confirm schedule next visit.

Two weeks after visit 0, the subject will return to the research center, where a new measurement of the electrical, photometric and colorimetric variables as well as self-assessment of oily skin, a standardized photograph with visual assessment and self-image questionnaire is made. This procedure is repeated by the 4th week, additionally, the subject will answer the last part of the perception survey in this visit. Once this is completed the product application phase will be terminated and the amount of remaining product as well as any significant journal entries will be registered at this point.

Throughout the study there will be tolerance and safety monitoring in every visit and follow-up call, as follows: Upon first application of the investigational product there will be an observation of the subject during a 15-minute period done by the research staff, a physician will be available to assess any possible allergic reaction or significant irritation.

The research staff will examine the application site of the research product to find potential local reactions and will ask about any systemic symptom. If no adverse reactions occur, the information will be recorded. Similarly, if any adverse reaction, systemic reaction or adverse event occurs it will be recorded and the physician will take the necessary measures to ensure subject safety according to his expert judgement and initiate event reporting according to applicable regulation. Finally, in every phone call made by the call center, adherence and tolerance questions will be made and recorded.

At the 5th week, the subject will receive a final follow-up call to record any events that might have appeared after removing the product, thus ending follow-up phase

ELIGIBILITY:
Eligibility criteria Healthy adult men and women with oily skin from the municipality of Chia and neighboring communities.

Inclusion criteria:

* Adult (i.e., over 18 years old) men or women.
* Oily or acne-prone skin as defined by self-assessment
* Accepts and signs the informed consent.

Exclusion criteria

* Pregnant or breast-feeding women
* Subjects with a chronic disease that requires medication
* Subjects with known diagnosis of cancer
* Smoking habit or alcohol consumption habit (i.e., once a day or more)
* Recreational or medicinal use of cannabinoids
* Skin diseases (i.e., diseases that require care of a dermatologist)
* Current medication uses such as: Immunomodulators, antibiotics, corticoids or retinoids
* Hypersensitivity to any component of the research product
* Involvement in other clinical or cosmetic studies in the last 6 months
* Recent exposure to sun causing sun tanning (i.e., as reported by the subject causing discomfort or change in the usual appearance of the skin)
* Permanent decoration of the skin in the test area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect on hydration of a single application of the topical preparation on facial skin | Change from baseline at 1 and 3 hours
  Evaluate the effect on hydration of a single application of the topical preparation on facial skin, through the direct measurement of its electrical properties as an indicator of water content at 1 and 3 hours. Measurement of the water content of the stratum corneum by capacitance.
Evaluate the effect on hydration of periodic application of the topical preparation on facial skin | Change from baseline at 2 and 4 weeks
  Evaluate the effect on hydration of periodic application of the topical preparation on facial skin, through the direct measurement of its electrical properties as an indicator of water content at 2 and 4 weeks. Measurement of the water content of the stratum corneum by capacitance.

SECONDARY OUTCOMES:
Evaluate the short-term change in instrumentally assessed measurement of oily skin | Change from baseline at 1 and 3 hours
  Evaluate the short-term change in instrumentally assessed measurement of oily skin (i.e., 1 and 3 hours), through photometrical transparency change of a translucent plastic strip.
Evaluate the long-term change in instrumentally assessed measurement of oily skin | Change from baseline at 2 and 4 weeks
  Evaluate the long-term change in instrumentally assessed measurement of oily skin (i.e., 2 and 4 weeks), through photometrical transparency change of a translucent plastic strip.
Evaluate the short-term change in instrumentally measured skin biochromophores | Change from baseline at 1 and 3 hours
  Evaluate the short-term change in instrumentally measured skin biochromophores (i.e., 1 and 3 hours)
Evaluate the long-term change in instrumentally measured skin biochromophores | Change from baseline at 2 and 4 weeks
  Evaluate the long-term change in instrumentally measured skin biochromophores (i.e., 2 and 4 weeks)
Evaluate the short-term effect (i.e., 1 and 3 hours) of this topical preparation on subjective assessment of oily skin | Change from baseline at 1 and 3 hours
  Evaluate the short-term effect (i.e., 1 and 3 hours) of this topical preparation on subjective assessment of oily skin, through the application of a validated questionnaire. Subjects will evaluate the degree of oiliness in a visual analog scale of 0 to 10 (i.e., 0: normal skin; 10: very severe oiliness)
Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on subjective assessment of oily skin | Change from baseline at 2 and 4 weeks
  Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on subjective assessment of oily skin, through the application of a validated questionnaire Subjects will evaluate the degree of oiliness in a visual analog scale of 0 to 10 (i.e., 0: normal skin; 10: very severe oiliness)
Evaluate the short-term effect (i.e., 1 and 3 hours) of this topical preparation on the skin appearance | Change from baseline at 1 and 3 hours
  Evaluate the short-term effect (i.e., 1 and 3 hours) of this topical preparation on the skin appearance, trough standardized photography and investigator evaluation. Subjects will be assessed by the investigation staff in comparison with baseline as follows: Almost clear if 90-99% clearance is observed Marked improvement if 75-89% clearance is observed Moderate improvement if 50-74% clearance is observed Minimal improvement if 25-49% clearance is observed No change if 0-24% clearance from baseline is observed
Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on the skin appearance | Change from baseline at 2 and 4 weeks
  Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on the skin appearance, trough standardized photography and investigator evaluation. Subjects will be assessed by the investigation staff in comparison with baseline as follows: Almost clear if 90-99% clearance is observed Marked improvement if 75-89% clearance is observed Moderate improvement if 50-74% clearance is observed Minimal improvement if 25-49% clearance is observed No change if 0-24% clearance from baseline is observed
Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on quality of life | Change from baseline at 2 and 4 weeks
  Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on quality of life, through the application of a standardized self-image questionnaire. The OSSIQ questionnaire will be used to perform self-image assessment by the subject using a five-point scale (never 0, rarely 1, sometimes 2, often 3, and always 4) to score 18 questions.
Evaluate the short and long-term emollient effect and acceptance of this topical preparation | 0 hours, 1 hour, and 4 weeks
  Evaluate the short and long-term emollient effect and acceptance of this topical preparation, through the application of a perception survey (i.e., 0 hours, 1 hours and 4 weeks). Perceived skinfeel attributes of creams and lotions (appearance, rub-in, absorption, appearance of skin, immediate and delayed after-feel) have been evaluated using a trained descriptive panel. In previously published studies researchers used the skinfeel spectrum descriptive analysis method to characterize skin care products. They used strict protocols for manipulation and precisely defined terms to describe the qualitative properties and their relative intensities in each product. The evaluation process was divided into four categories: pick-up (i.e., firmness, stickiness, cohesiveness, peaking); rub-out (i.e., wetness, spreadability, thickness, absorbency); residual feel; and appearance, immediate and after 20 minutes (i.e., glossy, sticky, slippery, oily, waxy, greasy
Evaluate the short and long-term tolerance of this topical preparation | 0 hours, 1 hour, and 4 weeks
  Evaluate the short and long-term tolerance of this topical preparation, through the application of a perception survey. This is scored by investigators using a four-point scale: absent, mild, moderate and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Granados, MD., MSc., Principal Investigator — Centro de Atencion e Investigacion Medica
Locations (1):
- VITA, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapoor S, Saraf S. Assessment of viscoelasticity and hydration effect of herbal moisturizers using bioengineering techniques. Pharmacogn Mag. 2010 Oct;6(24):298-304. doi: 10.4103/0973-1296.71797. PMID 21120032
- [Background] Poli F, Dreno B, Verschoore M. An epidemiological study of acne in female adults: results of a survey conducted in France. J Eur Acad Dermatol Venereol. 2001 Nov;15(6):541-5. doi: 10.1046/j.1468-3083.2001.00357.x. PMID 11843213
- [Background] Arbuckle R, Clark M, Harness J, Bonner N, Scott J, Draelos Z, Rizer R, Yeh Y, Copley-Merriman K. Item reduction and psychometric validation of the Oily Skin Self Assessment Scale (OSSAS) and the Oily Skin Impact Scale (OSIS). Value Health. 2009 Jul-Aug;12(5):828-37. doi: 10.1111/j.1524-4733.2009.00504.x. PMID 19508666
- [Background] Segot-Chicq E, Compan-Zaouati D, Wolkenstein P, Consoli S, Rodary C, Delvigne V, Guillou V, Poli F. Development and validation of a questionnaire to evaluate how a cosmetic product for oily skin is able to improve well-being in women. J Eur Acad Dermatol Venereol. 2007 Oct;21(9):1181-6. doi: 10.1111/j.1468-3083.2007.02193.x. PMID 17894702
- [Background] Biro T, Toth BI, Hasko G, Paus R, Pacher P. The endocannabinoid system of the skin in health and disease: novel perspectives and therapeutic opportunities. Trends Pharmacol Sci. 2009 Aug;30(8):411-20. doi: 10.1016/j.tips.2009.05.004. Epub 2009 Jul 14. PMID 19608284
- [Background] Kupczyk P, Reich A, Szepietowski JC. Cannabinoid system in the skin - a possible target for future therapies in dermatology. Exp Dermatol. 2009 Aug;18(8):669-79. doi: 10.1111/j.1600-0625.2009.00923.x. PMID 19664006
- [Background] Citti C, Pacchetti B, Vandelli MA, Forni F, Cannazza G. Analysis of cannabinoids in commercial hemp seed oil and decarboxylation kinetics studies of cannabidiolic acid (CBDA). J Pharm Biomed Anal. 2018 Feb 5;149:532-540. doi: 10.1016/j.jpba.2017.11.044. Epub 2017 Nov 20. PMID 29182999
- [Background] Mikulcova V, Kasparkova V, Humpolicek P, Bunkova L. Formulation, Characterization and Properties of Hemp Seed Oil and Its Emulsions. Molecules. 2017 Apr 27;22(5):700. doi: 10.3390/molecules22050700. PMID 28448475
- [Background] Eccles M, Grimshaw J, Campbell M, Ramsay C. Research designs for studies evaluating the effectiveness of change and improvement strategies. Qual Saf Health Care. 2003 Feb;12(1):47-52. doi: 10.1136/qhc.12.1.47. PMID 12571345
- [Background] Tsai TH, Chuang LT, Lien TJ, Liing YR, Chen WY, Tsai PJ. Rosmarinus officinalis extract suppresses Propionibacterium acnes-induced inflammatory responses. J Med Food. 2013 Apr;16(4):324-33. doi: 10.1089/jmf.2012.2577. Epub 2013 Mar 20. PMID 23514231
- [Background] Rawlings AV, Canestrari DA, Dobkowski B. Moisturizer technology versus clinical performance. Dermatol Ther. 2004;17 Suppl 1:49-56. doi: 10.1111/j.1396-0296.2004.04s1006.x. PMID 14728699
- [Background] Petry T, Bury D, Fautz R, Hauser M, Huber B, Markowetz A, Mishra S, Rettinger K, Schuh W, Teichert T. Review of data on the dermal penetration of mineral oils and waxes used in cosmetic applications. Toxicol Lett. 2017 Oct 5;280:70-78. doi: 10.1016/j.toxlet.2017.07.899. Epub 2017 Aug 5. PMID 28789996
- [Background] Reuter J, Merfort I, Schempp CM. Botanicals in dermatology: an evidence-based review. Am J Clin Dermatol. 2010;11(4):247-67. doi: 10.2165/11533220-000000000-00000. PMID 20509719
- [Background] Iffland K, Grotenhermen F. An Update on Safety and Side Effects of Cannabidiol: A Review of Clinical Data and Relevant Animal Studies. Cannabis Cannabinoid Res. 2017 Jun 1;2(1):139-154. doi: 10.1089/can.2016.0034. eCollection 2017. PMID 28861514
- [Background] Darlenski R, Sassning S, Tsankov N, Fluhr JW. Non-invasive in vivo methods for investigation of the skin barrier physical properties. Eur J Pharm Biopharm. 2009 Jun;72(2):295-303. doi: 10.1016/j.ejpb.2008.11.013. Epub 2008 Dec 11. PMID 19118626
- [Background] Loden M. The clinical benefit of moisturizers. J Eur Acad Dermatol Venereol. 2005 Nov;19(6):672-88; quiz 686-7. doi: 10.1111/j.1468-3083.2005.01326.x. PMID 16268870
- [Background] Parente ME, Gambaro A, Solana G. Study of sensory properties of emollients used in cosmetics and their correlation with physicochemical properties. J Cosmet Sci. 2005 May-Jun;56(3):175-82. PMID 16116522
- [Background] Lukic M, Jaksic I, Krstonosic V, Cekic N, Savic S. A combined approach in characterization of an effective w/o hand cream: the influence of emollient on textural, sensorial and in vivo skin performance. Int J Cosmet Sci. 2012 Apr;34(2):140-9. doi: 10.1111/j.1468-2494.2011.00693.x. Epub 2011 Dec 6. PMID 22085371